CLINICAL TRIAL: NCT06085456
Title: Individualized Health Management of Epithelial Ovarian Cancer: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2023-0202
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Diagnosis; Prognosis
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EOC group: Patients diagnosed with epithelial ovarian cancer
  Interventions: Diagnostic Test: Hematologic features
- Control group: Patients diagnosed with benign gynecological diseases, including ovarian cysts, uterine fibroids and uterine prolapse.
  Interventions: Diagnostic Test: Hematologic features

INTERVENTIONS:
Diagnostic Test: Hematologic features — Hematologic features including blood routine tests, blood biochemical indicators, and tumor markers before surgery

SUMMARY:
The purpose of this study is to identify the demographic and sociological characteristics of epithelial ovarian cancer in a cohort, identify the risk factors of epithelial ovarian cancer, effectively identify the high-risk population of epithelial ovarian cancer in the population, implement standardized health management, and clarify the effect of standardized health management on the incidence and prognosis of epithelial ovarian cancer. It can also provide a case control population for the clinical cohort of epithelial ovarian cancer to benefit the majority of postoperative patients.

DETAILED DESCRIPTION:
1. The clinical characteristics, preoperative hematological parameters of patients with epithelial ovarian cancer and patients with benign gynecological diseases, and the pathological stage, grade and features extracted by PET/CT images of patients with epithelial ovarian cancer were recorded.
2. Patients from Renji Hospital were divided into training group and test group at a ratio of 7:3, and patients from Shanghai First Maternity and Infant Hospital were used as external validation group.
3. The training group was used to establish the diagnosis and prognosis prediction model of epithelial ovarian cancer, and the test group and the external validation group were used to verify the model, and the area under the ROC curve, accuracy, specificity, and sensitivity were used to evaluate the effect of the model.
4. For machine learning models, SHAP and LIME algorithms were used for model interpretation.
5. Unsupervised clustering algorithm was used to distinguish the subgroups of epithelial ovarian cancer patients, and KM was used to analyze the overall survival (OS) and progression-free survival (PFS) to predict the survival and recurrence of the subgroups. Overall survival (OS) was defined as the time from the first diagnosis of epithelial ovarian cancer to the confirmation of death or the end of follow-up. Progression-free survival (PFS) was defined as the time from the first diagnosis of epithelial ovarian cancer to the confirmation of disease progression or the end of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as primary epithelial ovarian cancer with definite pathological stage and grade and underwent preoperative PET/CT examination, or patients diagnosed as benign gynecological diseases including ovarian cysts, uterine fibroids, and uterine prolapse.
* age between 18 to 80 years old;
* complete preoperative blood routine test results, blood biochemical indicators, and tumor markers;

Exclusion Criteria:

* complicated with acute or chronic genital tract infectious diseases;
* patients with diagnosed tumors other than ovarian cancer;
* complicated with severe systemic diseases;
* pregnant or lactating women;
* patients diagnosed with recurrent epithelial ovarian cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as primary epithelial ovarian cancer or patients diagnosed as benign gynecological diseases including ovarian cysts, uterine fibroids, and uterine prolapse
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of diagnosed patients | one month after surgery
  Patients were diagnosed with epithelial ovarian cancer or benign gynecological diseases (including ovarian cysts, uterine fibroids, and uterine prolapse). The blood characteristics of patients with epithelial ovarian cancer and patients with benign gynecological diseases (including ovarian cysts, uterine fibroids, and uterine prolapse) were compared to observe the performance of the study model in predicting disease diagnosis

SECONDARY OUTCOMES:
Overall survival | up to 5 years
  The time from the first surgical or biopsy diagnosis of epithelial ovarian cancer to confirmed death or the end of follow-up
Progression-free survival | up to 5 years
  The time from the first surgical or needle biopsy diagnosis of epithelial ovarian cancer to the confirmation of disease progression or the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Zhao, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No